CLINICAL TRIAL: NCT06641102
Title: Healing Track Randomized Clinical Trial
Brief Title: Healing Track Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Healing Track (Unknown)
Responsible Party: Principal Investigator, David Putrino, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-24-00080
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Chronic Back Pain
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study team will remain unblinded for study procedures. Statistical analysis will be performed by a statistician who is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Participants with Chronic Back Pain in Self-Guided Program (Experimental): Participants with CBP in a self-guided program that includes videos, guided meditations, and worksheets that are delivered to users in 10 different topical modules.
  Interventions: Other: Self-Guided Program (Tier 1)
- Participants with Chronic Back Pain in Coach Assisted Program (Experimental): Participants with CBP in a one-on-one coaching program that sets users up with trained PRT coaches who will walk them through the program individually.
  Interventions: Other: Coach Assisted Program (Tier 3)
- Participants receiving Standard of Care (Active Comparator): Standard of care (SOC) control group in adults with CBP.
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Other: Self-Guided Program (Tier 1) — The study intervention is a smartphone application.
  Tier 1: self-guided program, includes videos, guided meditations, and worksheets that are delivered to users in 10 different topical modules. Two modules are delivered per week, with email reminders. It will emphasize that PRT is a practice that requires users to come back to the material regularly to help retrain the brain often (just like how you need to practice and complete exercises between PT sessions).
  Arms: Participants with Chronic Back Pain in Self-Guided Program
Other: Coach Assisted Program (Tier 3) — The study intervention is a smartphone application.
  Tier 3: one-on-one coaching program that sets users up with trained PRT coaches who will walk them through the program individually. Users will meet with the assigned coaches once per week for an hour-long Zoom-hosted session that covers the same information as Tier 1, however in a completely personal and individualized way, focusing on the content that is most relevant for the user/patient at the time of the session. Tier 3 users will also receive materials from their coaches (e.g. videos, meditations, etc.) to support their own practice between session.
  Arms: Participants with Chronic Back Pain in Coach Assisted Program
Other: Standard of Care (SOC) — SOC is defined as a comprehensive clinical care plan, including a consultation with physiatrist and prescribed interventions, which will capture a comparison representative of all potential interventions that are recommended for an individual.
  Arms: Participants receiving Standard of Care

SUMMARY:
This is a randomized clinical trial to evaluate a digital pain reprocessing therapy (PRT) intervention for chronic back pain (CBP).

The purpose of this research is to test whether a new digital treatment for chronic pain works as well as traditional treatments for chronic back pain (CBP). Some people with CBP experienced side effects from other treatments, or previous treatments did not relieve pain, so this research aims to see if a digital therapy is a better option for CBP.

This study will assess changes in pain intensity from PRT intervention compared to a standard of care (SOC) control group in adults with CBP. SOC is defined as a comprehensive clinical care plan, including a consultation with physiatrist and prescribed interventions, which will capture a comparison representative of all potential interventions that are recommended for an individual.

The research team plans to enroll 180 participants who will be randomized into one of three groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 70
* Chronic Back Pain- CBP will be defined according to the criteria established by a recent NIH task force
* Pain duration must be at least 3 months, with back pain being an ongoing problem for at least half the days of the last 6 months. That is, patients can meet criteria by either reporting pain every day for the past 3 months, or by reporting pain on half or more of the days for the past 6+ months.
* Patients must rate pain intensity at 4/10 or greater on the Brief Pain Inventory-Short Form (BPISF) (on the item measuring average pain over the last week).
* Participants must also be comfortable and able to communicate via email or text message, as several study measures are collected in this manner.
* Able to use a smartphone

Exclusion Criteria:

* Back pain associated with compensation or litigation issues as determined by self-report within the past year
* Leg pain is greater than back pain, as this suggests neuropathic pain, which may be less responsive to psychotherapy
* Cauda Equina syndrome, as screened for by self-reported inability to control bowel or bladder function
* Self-reported diagnoses of schizophrenia, multiple personality disorder, or dissociative identity disorder
* Self-reported use of intravenous drugs, due to concerns about infections and subject compliance with experimental protocols

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory Short Form | <Day 0, Day 0, Day 1, Week 6, Week 10, Month 8.5
  A 9-item instrument with total score from 0 to 10, with higher score indicating worse outcomes. Full scale from 0 to 10, with higher score indicating more pain symptoms.
  Minimum score: 0 (no pain) Maximum score: 10 (pain as bad as you can imagine)

CONTACTS AND LOCATIONS:
Overall Officials: David Putrino, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai - Abilities Research Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.